CLINICAL TRIAL: NCT01080690
Title: Endosonography For Right Side Acute Intestinal Mal-Symptoms (EFRAIM- Study)
Acronym: EFRAIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Prof. A. Meining, TUM, Technical University Munich
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 01102
Record Dates: First submitted 2010-01-27; First posted 2010-03-04 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2010-02

CONDITIONS: Abdominal Pain
Keywords: endosonography, right side abdominal pain; Endosonography (diagnostic value in right side abdominal pain)
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EGD (Active Comparator): In this arm EGD will be performed before EUS
  Interventions: Procedure: EGD
- EUS (Active Comparator): In this arm, EUS will be performed before EGD.
  Interventions: Procedure: EUS

INTERVENTIONS:
Procedure: EGD — In this arm EGD will be performed before EUS.
  Other Names: EGD: A standard diagnostic EGD will be performed.; EUS: A standard diagnostic EUS will be performed.
  Arms: EGD
Procedure: EUS — In this arm EUS will be performed before EGD.
  Arms: EUS

SUMMARY:
Hypothesis: Endosonography (EUS) in a single setting is equivalent to the standard algorithm combining abdominal sonography, gastroscopy, endosonography in patients with acute right side abdominal pain.

Patients with acute right side abdominal pain will be randomized in one of two groups. In each group all examinations (sonography, gastroscopy, endosonography) will be performed. The study group only defines the order of the examinations. Abdominal sonography will always be performed before endoscopic procedures. In group 1, gastroscopy is first followed by endosonography. In group 2 endosonography is first followed by gastroscopy.

Two physicians will review all results of all examinations, patient charts as well as a follow up visit and establish a clinical diagnosis.

Yield of the clinical diagnosis by EUS results alone will be compared to the yield by combined results of sonography, EGD and EUS.

ELIGIBILITY:
Inclusion Criteria:

* acute right side abdominal pain
* willing participate study

Exclusion Criteria:

* acute disease
* malignancy
* other disease which might cause discomfort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Yield of the clinical diagnosis by EUS results alone will be compared to the yield by combined results of sonography, EGD and EUS. | within the first week of complaints

SECONDARY OUTCOMES:
Calculate the time and cost savings and number of procedures for endosonography alone versus the combined approach of abd. sonography, gastroscopy and endosonography. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Meining, Prof., Principal Investigator — II Med Dep, TU Munich
Locations (1):
- Klinikum r.d. Isar, Technical University Munich, Munich, Germany